CLINICAL TRIAL: NCT00048802
Title: Treatment and Outcome of Early Onset Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH060845 (NIH); R01MH060845 (NIH); DSIR 84-CTM
Record Dates: First submitted 2002-11-08; First posted 2002-11-13 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Bipolar Disorder
Keywords: Adolescence
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium; Olanzapine; Valproic Acid; Risperidone; Quetiapine Fumarate; ziprasidone

INTERVENTIONS:
Drug: Lithium
Drug: Olanzapine
Drug: Divalproex
Drug: Risperidone
Drug: Quetiapine
Drug: Ziprasidone
Drug: Aripriprazole

SUMMARY:
This study will compare the effectiveness in the maintenance of continuing adjunctive atypical antipsychotic medication compared to traditional mood stabilizer(s) alone in the maintenance treatment of adolescents with bipolar disorder.

DETAILED DESCRIPTION:
In children and adolescents, bipolar disorder is often accompanied by symptoms such as hallucinations, delusions, or paranoia that require acute treatment with a combination of an atypical antipsychotic medication and a mood stabilizer. It is not known if it is necessary to continue treatment with the atypical antipsychotic medication after the child's symptoms have remitted.

Participants in this study are treated with lithium, divalproex (Depakote), and one of the following atypical antipsychotic medications: olanzapine (Zyprexa), risperidone (Risperdal) or quetiapine (Seroquel) for at least 24 weeks. Participants who have already begun combination therapy with at least one of the mood stabilizers and atypical antipsychotic medications listed above are also encouraged to enroll in this study. After participants have been on combination therapy for at least 24 weeks they will then be randomly assigned to one of two groups. The first group will continue to receive active mood stabilizer and atypical antipsychotic medication. The second group will receive active mood stabilizer and placebo. Participants are assessed weekly and followed for up to 18 months.

ELIGIBILITY:
Inclusion criteria:

* Have a diagnosis of Bipolar I Disorder;
* Have had aggressive and/or psychotic features (delusions, hallucinations and/or thought disorder) during the most recent manic episode;
* Is willing to be treated or is already being treated with the combination of mood stabilizer(s) (lithium or Depakote) and an atypical antipsychotic medication (Abilify, Geodon, Risperdal, Seroquel, or Zyprexa);
* Live in the NY Metropolitan area;
* Able to attend weekly to biweekly office visits

Exclusion Criteria:

* Medical contraindication to treatment with lithium and divalproex
* Seizure disorder
* Pregnancy
* Unwillingness to use acceptable methods of birth control if sexually active
* IQ less than 70
* Substance-induced mood disorder or mood disorder due to a general medical condition
* Prior experience with re-emergence of psychotic features or severe aggression within 6 months of antipsychotic medication discontinuation under circumstances similar to those in the study
* Potentially lethal suicide attempts or infliction of serious injury upon someone during most severe bipolar episode
* High risk for running away or truancy

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2002-08; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Zucker Hillside Hospital, Long Island Jewish Medical Center, Glen Oaks, New York, United States

REFERENCES:
- [Background] Kafantaris V, Coletti DJ, Dicker R, Padula G, Kane JM. Adjunctive antipsychotic treatment of adolescents with bipolar psychosis. J Am Acad Child Adolesc Psychiatry. 2001 Dec;40(12):1448-56. doi: 10.1097/00004583-200112000-00016. PMID 11765291
- [Background] Kafantaris V. Treatment of bipolar disorder in children and adolescents. J Am Acad Child Adolesc Psychiatry. 1995 Jun;34(6):732-41. doi: 10.1097/00004583-199506000-00013. PMID 7608046
- [Background] Kafantaris V, Coletti D, Dicker R, Padula G, Kane JM. Lithium treatment of acute mania in adolescents: a large open trial. J Am Acad Child Adolesc Psychiatry. 2003 Sep;42(9):1038-45. doi: 10.1097/01.CHI.0000070247.24125.24. PMID 12960703